CLINICAL TRIAL: NCT01761331
Title: Acupuncture in Infantile Colic - a Three Armed Randomized Multi Center Trial Comparing Acupuncture in a Standardized Point, Acupuncture in Individually Chosen Points and no Acupuncture
Brief Title: Acupuncture in Infantile Colic - a Three Armed Randomized Multi Center Trial (ACU-COL)
Acronym: ACU-COL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Ekhagastiftelsen (Other)
Responsible Party: Principal Investigator, Kajsa Landgren, Principal Investigator, Lund University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LU-HSC-KL2013
Record Dates: First submitted 2012-12-29; First posted 2013-01-04 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Infantile Colic
Keywords: infant, colic, crying, acupuncture, stooling, sleep
MeSH Terms: conditions — Colic; Crying | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A: Standardized acupuncture (Active Comparator): Infants come to the clinic twice a week for three weeks. Parents meet a nurse and hand the infant to her. The nurse brings the infant to a room where another nurse, trained in acupuncture, is alone with the infant for five minutes. Intervention: Infants in the standardized acupuncture group get minimal acupuncture: one needle is inserted about 3 mm in the point LI4 on the infants hands, unilaterally, for 2-10 seconds and then withdrawn.
  Interventions: Other: Acupuncture
- Group B: Individualized acupuncture (Active Comparator): Infants come to the clinic twice a week for three weeks. Parents meet a nurse and hand the infant to her. The nurse brings the infant to a room where another nurse, trained in acupuncture, is alone with the infant for five minutes. Infants in the individualized acupuncture group get acupuncture in points chosen by the acupuncturists according to symptoms: maximum 5 needles are inserted about 3 mm in points recommended in a guideline produced for the trial. Needles are retained for maximum one minute.
  Interventions: Other: Acupuncture
- Group C: No acupuncture (No Intervention): Infants come to the clinic twice a week for three weeks. Parents meet a nurse and hand the infant to her. The nurse brings the infant to a room where another nurse, trained in acupuncture, is alone with the infant for five minutes. The nurse hold the infant´s hand and talks to it but no acupuncture is given.

INTERVENTIONS:
Other: Acupuncture — Minimal standardized acupuncture: one needle is inserted about 3 mm in the point LI4 on the infants hands, unilaterally, for 2-10 seconds and then withdrawn.
  Individualized acupuncture: maximum 5 needles are inserted, about 3 mm deep, in points chosen by the acupuncturists according to symptoms, in points recommended in a guideline produced for the trial. Needles are retained for maximum one minute.
  Arms: Group A: Standardized acupuncture; Group B: Individualized acupuncture

SUMMARY:
The purpose of this prospective randomized three armed, multi center study is to compare the effect of two types of acupuncture and no acupuncture in 2-8 weeks old infants with infantile colic. Group A will get standardized minimal acupuncture in LI4, group B will get individualized acupuncture in different points according to symptoms and group C will not get acupuncture. Parents (who register the infants crying) and the nurse they meet at the study CHC are blinded.

DETAILED DESCRIPTION:
Infantile colic is a common problem, affecting 10-20% of newborns. Both the baby and the parents are suffering and there is a risk that the early relationship is disturbed. There is no safe and effective drug and the use of complementary medicine is increasing in spite of weak or no evidence. Acupuncture releases different neurotransmitters and hormones, is calming, gives pain reduction and affects digestion. Therefore it is reasonable that acupuncture can have effect in colic. Acupuncture in infantile colic has shown promising results in the few scientific trials conducted. These trials have evaluated the effect of standardized minimal acupuncture in the acupuncture points Large Intestine 4 (LI4) (two trials) or Stomach 36 (ST36) (one recent trial). In this prospective randomized three armed, multi center study performed at Child Health Centers in three towns, the effect of acupuncture in reducing symptoms in infants, 2-8 weeks old, with colic will be investigated. Two types of acupuncture: standardized minimal acupuncture in LI4 and individualized acupuncture in different points according to symptoms will be compared to an untreated group. Parents (who register the infants crying) and the nurse they meet at the study CHC are blinded.

Parents will get information about the trial from nurses and doctors at Child Health Centers (CHC) or from a web-site (www.spädbarnskolik.se). Parents who are interested in letting their infant participate in the trial get further information and sign informed consent. The trial is approved by the ethical board at Lund University.

Infant´s crying, fussing, sleep, feeding and stooling will be registered in a diary during a baseline week. Infants who cry/fuss more than three hours/day, more than three days during this week is included and randomized. Beside their ordinary contacts with their Child Health Center (CHC), infants and their parents are invited to visit a study CHC twice a week for two weeks, where they meet a nurse for about 20 minutes. Parents can describe their situation, discuss the infant´s symptoms and get advice. This nurse is blinded to which group the infant is randomized to. She carries the baby to another room and hands over the infant to a nurse, trained in acupuncture. The acupuncture nurse randomizes the infants to one of three groups, following a randomization list produced by the research department at Lund University Hospital. Group A will get standardized minimal acupuncture: one needle is inserted about 3 mm in the point LI4 on the infants hands, unilaterally, for 2-10 seconds and then withdrawn. Group B will get individualized acupuncture in points chosen by the acupuncturists according to symptoms: maximum 5 needles are inserted about 3 mm in points recommended in a guideline produced for the trial after discussions with experienced pediatric acupuncturists. Needles are retained for maximum one minute. Group C will not get acupuncture but will otherwise be treated similarly: they will be with the acupuncture nurse for five minutes while she holds the hand of the baby and talks to it in a calm voice. The acupuncture nurse make notes about bleeding and other possible side effects, and if the baby is crying. After approximately five minutes the acupuncture nurse calls the study nurse who carries the baby back to the parents. At every visit the study nurse asks parents if they have noticed any side effects, and asks if parents believe their baby gets acupuncture or not.

During the two intervention weeks and one week after the last visit to the study CHC parents register the infants behavior daily in a diary. Statistical analyses will be made from the diaries.

ELIGIBILITY:
Inclusion Criteria:

* otherwise healthy infants
* crying/fussing more than three hours/day more than three days in the same week
* has tried cow´s milk protein free diet for at least five days

Exclusion Criteria:

* born before week 36
* has tried acupuncture treatment
* dont gain weight properly
* taking other medicine than dimethicone or lactobacillus reuteri
* parents who don´t understand Swedish

Ages: 2 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
change in crying | mean values for crying during the baseline week, during each of the two intervention weeks and during the week after the last treatment
  Difference over time and between groups in reduction in % of colicky crying, crying and fussing in minutes/day

SECONDARY OUTCOMES:
change in stooling | mean values for stooling during the baseline week, during each of the two intervention weeks and during the week after the last treatment
  The frequency of stooling per day

OTHER OUTCOMES:
Change in hours of sleep | mean values for sleep and length of undisturbed sleep during the baseline week, during each of the two intervention weeks and during the week after the last treatment
  Hours of sleep per day
side effects | each of the four visits to the study CHC and one week after the last visit
  At each visit parents will be asked by the study nurse whether they have noticed any side effects that they believe can be associated with acupuncture. One week after the last visit they will, by telephone, be asked the same question by the study coordinator.
Blinding | each of the four visits to the study CHC and one week after the last visit
  At each visit parents will be asked by the study nurse whether they believe that their infant is allocated to acupuncture or not. One week after the last visit they will, by telephone, be asked the same question by the study coordinator.

CONTACTS AND LOCATIONS:
Overall Officials: Kajsa Landgren, PhD, Principal Investigator — Lund University
Locations (4):
- Sweden (4):
  - Arlöv vårdcentral, BVC, Arlöv, Skåne County
  - Askims vårdcentral, BVC, Askim, Västra Götaland County
  - Tullgårdens BVC, Karlskrona
  - Valla Vårdcentral, BVC, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Landgren K, Hallstrom I, Tiberg I. The effect of two types of minimal acupuncture on stooling, sleeping and feeding in infants with colic: secondary analysis of a multicentre RCT in Sweden (ACU-COL). Acupunct Med. 2021 Apr;39(2):106-115. doi: 10.1177/0964528420920308. Epub 2020 May 6. PMID 32375501
- [Derived] Landgren K, Hallstrom I. Effect of minimal acupuncture for infantile colic: a multicentre, three-armed, single-blind, randomised controlled trial (ACU-COL). Acupunct Med. 2017 Jun;35(3):171-179. doi: 10.1136/acupmed-2016-011208. Epub 2017 Jan 16. PMID 28093383
- [Derived] Landgren K, Tiberg I, Hallstrom I. Standardized minimal acupuncture, individualized acupuncture, and no acupuncture for infantile colic: study protocol for a multicenter randomized controlled trial - ACU-COL. BMC Complement Altern Med. 2015 Sep 14;15:325. doi: 10.1186/s12906-015-0850-x. PMID 26370560